CLINICAL TRIAL: NCT03448666
Title: A Phase II, Multicentric, Open Label, Non-randomized, Interventional Study of Pembrolizumab in Combination With Electrochemotherapy in Patients With Unresectable Melanoma With Superficial or Superficial and Visceral Metastases
Brief Title: ECT-Pembrolizumab in Patients With Unresectable Melanoma With Superficial or Superficial and Visceral Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no financial support
Sponsor: European Institute of Oncology (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 523
Record Dates: First submitted 2017-11-24; First posted 2018-02-28 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-06

CONDITIONS: Malignant Melanoma
Keywords: ECT; pembrolizumab; advanced melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Electrochemotherapy

STUDY DESIGN:
Intervention Model Description: This is a single arm trial with a single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab and elettrochemiotherapy (Experimental): drug: Pembrolizumab 200 mg flat dose every three weeks procedure: elettrochemiotherapy once after first pembrolizumab dose
  Interventions: Combination Product: Pembrolizumab

INTERVENTIONS:
Combination Product: Pembrolizumab — Electrochemotherapy will be performed with the CLINIPORATOR™ after the first treatment of Pembrolizumab
  Other Names: Electrochemotherapy

SUMMARY:
This is a Phase 2 multicenter, open label, non-randomized, interventional study enrolling 53 patients.The objectives and purposes of the clinical study described herein are to determine if concomitant Pembrolizumab (Keytruda) and ECT treatments are safe and able to improve local and systemic response rates.ECT will be performed with the CLINIPORATOR and a single IV dose of Bleomycin

DETAILED DESCRIPTION:
ECT induces immunogenic cell death of cancer cells with a more efficient antigen presentation of tumor-derived antigens by APCs to T-cells, particularly CD8+ antigen-specific T cells. Anti-PD-1 mAb reverts T-cell exhaustion induced by PD-1/PD-L1 and PD-L2 engagement on CD8+ T cells. Moreover, it may also be beneficial in the priming phase of the antitumor immune responses, inducing long-lived tumor antigen-specific CD8+ T-cell effectors.

The main hypothesis is to establish if concomitant treatment of Pembrolizumab and ECT is able to lead to a 20% increase of the ORR using as a reference the proportion of success available in the literature for Pembrolizumab.

The investigators will perform a proteomic analysis of sera of treated patients, collected before and after treatments, with particular emphasis on cytokines and chemokines, to evaluate possible markers associated with a better clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically confirmed advanced melanoma stages III b/c or IV, with at least the following superficial lesions: 5 lesions if diameter < 1 cm or 3 lesions if diameter > 1 cm.
2. Could have received previous therapy included CT, antiCTLA4 or antiBRAF/antiMEK treatment or be treatment naïve.
3. Be willing and able to provide written informed consent/assent for the trial.
4. Be >= 18 years of age on day of signing informed consent.
5. Have measurable disease based on RECIST 1.1.
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
7. Have a performance status ≤ 2 on the ECOG Performance Scale. (Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.)
8. Demonstrate adequate organ function as defined in
9. Have a baseline total body CT scan (brain MRI if brain metastasis are suspected)

   1. Patients with brain metastasis are allowed to participate if previously treated and brain lesion stability or inactivity is demonstrated. Patients with a history of brain metastasis are required to have a pre-baseline brain MRI at least 60 days (2 months) before the Screening/Baseline visit (Visit 1) for comparison to the Screening (Visit 1) MRI. Patients for whom MRI is contraindicated will undergo head CT. Stable/inactive disease is determined by comparing the pre- baseline and screening/baseline MRI/CT results.
   2. Patients presenting with brain metastasis at Screening/Baseline who had no known previous brain involvement and who had no brain MRI/CT tests at least 60 days (2 months) before Screening/Baseline are considered screening failures and will be excluded from study enrollment.
10. Have cutaneous or subcutaneous metastases from melanoma that are accessible for the application of electric pulses using the single use, sterile CLINIPORATOR™ electrodes (5 lesions if diameter <1 cm or 3 lesions if diameter >1 cm). For patients presenting with more than 7 lesions, the lesions with the largest diameters that fall within the <10 to 30 mm size requirements will be considered "target" lesions for RECIST criteria and study purposes. The others will be recorded and monitored but will not considered as Target.
11. Have lesions clearly requiring palliative treatment [e.g., symptomatic (bleeding, draining, painful), disfiguring or causing distress to the patient].
12. A treatment-free period of three (3) weeks before enrolling in the study. NOTE: Patients receiving concomitant treatments for unrelated existing pathologies are eligible for enrollment.
13. Life expectancy > 3 months.
14. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
15. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
16. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment or has any ongoing treatment for melanoma or with any non-study anticancer therapy or immunosuppressive agent.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients or known allergies to Bleomycin.
5. Has received a cumulative lifetime dose of Bleomycin exceeding 250 mg/m2
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Patient has a history of a malignancy (other than the disease under treatment in the study) within 5 years prior to first study drug administration. This should exclude adequately treated Stage 1 or Stage 2 basal/squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or other in situ cancers. Shorter intervals can be considered after discussion with Merck.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has epilepsy.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of (no-infectious) pneumonitis that require steroids or current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. Has primary ocular melanoma
21. Non-cutaneous/subcutaneous symptomatic or rapidly progressive metastases
22. Cardiac arrhythmias [e.g., significant ventricular arrhythmia such as persistent ventricular tachycardia and/or ventricular fibrillation; severe conduction disorders as atrioventricular block 2 and 3, sinoatrial block]
23. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate, as Determined by RECIST v1.1 | Baseline up to disease progression or death due to any cause, whichever occurs first (up to approximately 60 months)
  CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Pier Fr Ferrucci, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- IEO Istituto Europeo di Oncologia, Milan, Italy

IPD SHARING:
Plan to Share IPD: No